CLINICAL TRIAL: NCT00278746
Title: An Effectiveness Trial Examining the Addition of Zinc to the Current Case Management Package of Diarrhea in a Primary Health Care Setting.
Brief Title: Addition of Zinc to the Current Case Management Package of Diarrhea in a Primary Health Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: Ministry of Science and Technology, India (Other Government); United Nations Children's Fund, Delhi (Unknown); World Health Organization (Other)
Responsible Party: Nita Bhandari, Society for Applied Studies, New Delhi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-5268/PID/20/198/2004
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Diarrhea; Mortality; Hospitalization
Keywords: zinc; diarrhea; cluster randomization; hospitalization
MeSH Terms: conditions — Diarrhea | interventions — Zinc; ORALIT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Zinc and ORS were promoted for treatment of diarrhea in underfive children
  Interventions: Drug: Zinc and ORS
- 2 (Other): Promoted routine management of diarrhea in underfive with ORS
  Interventions: Drug: ORS only

INTERVENTIONS:
Drug: Zinc and ORS — Government and private providers and village health workers were trained to prescribe zinc and ORS for use in diarrheal episodes in 1 month to 5 years old children in intervention communities
  Arms: 1
Drug: ORS only — Promoted routine management of diarrhea in underfive with ORS
  Arms: 2

SUMMARY:
Several studies have shown the beneficial effect of zinc treatment in acute diarrhea. There was a significant reduction in duration of the treated episodes and in their severity as measured by diarrheal stool output or frequency. Zinc is a potentially important immunomodulator or nutraceutical which may have great impact as therapeutic agent in conditions like diarrhea and pneumonia. The issue is whether and how zinc should be introduced in primary health care programs for treatment of acute diarrhea. A practical, sustainable intervention for introduction of zinc as treatment of acute diarrhoea in national programs is therefore required. This study aimed to address this issue.

DETAILED DESCRIPTION:
This cluster randomized trial aimed at evaluating in a community based controlled effectiveness trial whether addition of 2RDA zinc as a therapeutic modality to the current case management package for diarrhoea in children aged between 1 month and 5 years, delivered through existing channels at village level, resulted in reduction in care seeking from health care providers, antibiotic and other drug use and increase in ORS use rates.

The intervention was being implemented in 6 PHCs; 3 intervention and 3 control.

Based on the experience of a pilot study and the formative research findings, common sources visited by caregivers for care seeking during morbidity were identified. These sources were selected as channels in partnership with the local government, to distribute zinc strips and ORS packets in intervention sites and only ORS packets in control sites. These channels were physicians (at the PHC and private practitioners), the auxiliary nurse midwives (ANMs) and Anganwadi workers (AWWs) of the Integrated Child Development Services (ICDS) Scheme. All the channels were trained and supplies of zinc strips and ORS packets, and ORS packets only were distributed in each pair of PHC in intervention and control sites respectively. Recommendations were developed and translated into local vernacular. A poster, incorporating these recommendations and pictures of zinc strips and ORS packets, was designed and put up at various places in the intervention sites. For outcome measurements, cross sectional surveys were conducted at 6 monthly intervals.

Process evaluation activities, which included observations of different channels and exit interviews with mothers after they had visited a channel were conducted.

In the two groups, zinc was used in 36.5% and 59.8% diarrheal episodes and ORS in 34.8% and 59.2% episodes in the 4 weeks preceding interviews in intervention areas. In control areas, ORS was used in 7.8% and 9.8% episodes. Care seeking for diarrhea, prescription of drugs of unknown identity and antibiotics for diarrhea reduced in intervention communities.

The study demonstrated that an intervention to improve diarrhea management with ORS and zinc is feasible and highly acceptable in rural Indian communities. The resulting health benefits were substantial and accomplished with a reduction in the cost to families for diarrhea treatment from current practices.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 5 years with diarrhea

Exclusion Criteria:

* Illness requiring referral to hospital

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20032 (Actual)
Dates: Start 2005-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To evaluate in a community based controlled effectiveness trial whether addition of zinc as a therapeutic modality for diarrhea delivered through existing channels, including at village level to the current case management package for under-five children | 20 months (Jan 2005 to Sep 2006)
- Reduction in visits to health care providers for treatment of illness | 20 months (Jan 2005 to Sep 2006)
- Reduction in drug use; antibiotics and other drugs during diarrheal illnesses | 20 months (Jan 2005 to Sep 2006)
- Increase in ORS use during diarrhea in the intervention communities. | 20 months (Jan 2005 to Sep 2006)

SECONDARY OUTCOMES:
- Reduction in all cause hospitalizations | 20 months (Jan 2005 to Sep 2006)

CONTACTS AND LOCATIONS:
Overall Officials: Nita Bhandari, PhD, Principal Investigator — Society for Applied Studies
Locations (1):
- Society for Applied Studies, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Bhandari N, Mazumder S, Taneja S, Dube B, Agarwal RC, Mahalanabis D, Fontaine O, Black RE, Bhan MK. Effectiveness of zinc supplementation plus oral rehydration salts compared with oral rehydration salts alone as a treatment for acute diarrhea in a primary care setting: a cluster randomized trial. Pediatrics. 2008 May;121(5):e1279-85. doi: 10.1542/peds.2007-1939. PMID 18450870